CLINICAL TRIAL: NCT00613119
Title: PET Evaluation of Brain Peripheral Benzodiazepine Receptors Using [11C]PBR28 in Neurological Disorders
Brief Title: PET Evaluation of Brain Peripheral Benzodiazepine Receptors Using [11C]PBR28 in Frontotemporal Dementia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080066; 08-M-0066
Record Dates: First submitted 2008-02-10; First posted 2008-02-12 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-07-13

CONDITIONS: Frontotemporal Lobar Degeneration; Dementia
Keywords: Inflammation; Frontotemporal Dementia; Dementia; PBR28; PET Imaging
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Dementia; Inflammation; Frontotemporal Dementia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use positron emission tomography (PET) imaging to measure a receptor in the brain that is involved in inflammation. Certain neurological disorders, possibly including frontotemporal dementia (FTD), are associated with increased inflammation in the brain. This study may help elucidate the relationship between FTD and inflammation.

Patients with FTD and healthy volunteers who are 35 years of age or older may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram, and blood and urine tests.

Participants undergo the following procedures:

* Whole body PET scan: PET uses small amounts of a radioactive chemical called a tracer that labels active areas of the brain so the activity can be seen with a special camera. The tracer used in this study is [11C]PBR28. Before starting the scan, a catheter (plastic tube) is placed in a vein in the arm to inject the tracer. Pictures are taken for 1 hour. This short scan is done to determine if [11C]PBR28 binds to the subject s receptors, since a number of people do not have binding. Subjects who have binding continue with brain PET and MRI scans, described below.
* Brain PET imaging: Before starting the scan, a catheter is placed in a vein in the arm to inject the tracer,<TAB> and another catheter is placed in an artery in the wrist to obtain blood samples during the scan. The subject lies on the scanner bed. A special mask is fitted to the head and attached to the bed to help keep the person s head still during the scan so the images will be clear. An 8-minute transmission scan is done just before the tracer is injected to provide measures of the brain that are helpful in calculating information from subsequent scans. After the tracer is injected, pictures are taken for about 2.5 hours, while the subject lies still on the scanner bed.
* Blood and urine tests are done the day of and the day following each PET scan.
* Magnetic resonance imaging (MRI): An MRI scan is done within 1 year (before or after) of the PET scan. This procedure uses a magnetic field and radio waves to produce images of the brain. The subject lies on a table that is moved into the scanner (a tube-like device), wearing earplugs to muffle the noise of the machine during the scanning process. The test takes about 1 hour....

DETAILED DESCRIPTION:
Objective:

Abnormal immune responses and inflammatory mechanisms have been implicated in the pathogenesis of certain neurodegenerative diseases. Frontotemporal dementia (FTD) is a neurodegenerative disease characterized by focal atrophy of the frontal and temporal lobes. Evidence supports the presence of inflammation in FTD; however, the relationship between inflammation and FTD pathogenesis is poorly understood. In addition, there is evidence of inflammation in temporal lobe epilepsy (TLE), a condition characterized by seizures originating from the mesial temporal lobe.

In response to brain inflammation, microglia are activated and over-express the peripheral benzodiazepine receptor (PBR). In normal conditions, PBR is expressed in low numbers. Measuring PBR density can identify areas of brain inflammation, because activated microglial cells in these areas express more PBR than microglial cells in resting conditions. Positron emission tomography (PET) imaging can quantify PBR density in vivo using radioligands that bind to PBR sites. One PBR-specific radioligand, [11C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195), has been used to identify areas of brain inflammation in patients with FTD. Unfortunately, [11C]PK11195 has several limitations, such as low brain uptake and low specific signal. A recently developed radioligand, [11C]N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine (PBR28), has higher affinity than [11C]PK11195 for PBR. [11C]PBR28 has never been used to study inflammation in FTD.

To further study brain inflammation in dementia and TLE, we wish to include patients with Alzheimer disease (AD) and TLE.

Study population:

In this protocol, we wish to evaluate 20 patients with FTD, 50 100 patients with AD, 20 patients with TLE, and 30 55 healthy volunteers.

Design:

Subjects will undergo a dedicated brain PET with [11C]PBR28, as well as a brain MRI. In AD patients and controls, 11C PBR28 PET and MRI will then be repeated after an interval of one year but no more than 5 years.

Outcome measures:

Outcome measures will be the amount of 11C PBR28 binding in the brain in FTD patients, AD patients, TLE patients and in healthy controls. We will quantify the radioligand s brain uptake, washout, plasma clearance, and distribution volume using compartmental modeling. Distribution volume is proportional to the density of receptors and is equal to the ratio at equilibrium of uptake in brain to the concentration of parent radiotracer in plasma. 11C PBR28 binding will also be compared between baseline and follow-up scans to determine the change in binding related to evolution of AD pathology and that related to normal aging.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with a diagnosis of Alzheimer disease or frontotemporal dementia (FTD). FTD patients with or without motor involvement may be included. FTD patients with either the frontal variant (also known as the behavioral variant) or the language variant of FTD may be included. AD and FTD patients must either meet capacity criteria to consent to research, or be able to assign a surrogate decision-maker who is able to consent to research on the subject s behalf.
* TLE patients must have clinically documented partial seizures with consistent EEG evidence as defined by the 1981 International Classification of Epileptic Seizures, refractory to standard antiepileptic treatment for at least one year. This criterion will be established by preliminary screening in the NINDS Clinical Epilepsy Section outpatient clinic, and if necessary, inpatient video-EEG monitoring.
* Healthy volunteers.

EXCLUSION CRITERIA:

* Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure, including that from this protocol, would exceed the guidelines set by the Radiation Safety Committee (RSC).
* Pregnancy or breast feeding.
* Positive result on urine screen for illicit drugs.
* Subjects who cannot lie on their back for extended periods of time.
* History of neurological disease other than FTD or AD or TLE.
* TLE patients:

  1. with a known treatable seizure etiology such as neoplastic or infectious disease
  2. with an MRI finding consistent with a brain tumor, trauma or arterial-venous malformations
  3. with seizure activity within 24 hours prior to the study.
  4. not capable of giving an informed consent.
* Presence of ferromagnetic metal in the body or heart pacemaker.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-01-31; Study Completion 2017-07-13

PRIMARY OUTCOMES:
Outcome measures will be the amount of [11C]PBR28 binding in the brain in FTD patients and in healthy controls.

SECONDARY OUTCOMES:
We will quantify the radioligand's brain uptake, washout, plasma clearance, and distribution volume using compartmental modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aisen PS, Davis KL. Inflammatory mechanisms in Alzheimer's disease: implications for therapy. Am J Psychiatry. 1994 Aug;151(8):1105-13. doi: 10.1176/ajp.151.8.1105. PMID 7518651
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Baker M, Mackenzie IR, Pickering-Brown SM, Gass J, Rademakers R, Lindholm C, Snowden J, Adamson J, Sadovnick AD, Rollinson S, Cannon A, Dwosh E, Neary D, Melquist S, Richardson A, Dickson D, Berger Z, Eriksen J, Robinson T, Zehr C, Dickey CA, Crook R, McGowan E, Mann D, Boeve B, Feldman H, Hutton M. Mutations in progranulin cause tau-negative frontotemporal dementia linked to chromosome 17. Nature. 2006 Aug 24;442(7105):916-9. doi: 10.1038/nature05016. Epub 2006 Jul 16. PMID 16862116
- [Derived] Paul S, Gallagher E, Liow JS, Mabins S, Henry K, Zoghbi SS, Gunn RN, Kreisl WC, Richards EM, Zanotti-Fregonara P, Morse CL, Hong J, Kowalski A, Pike VW, Innis RB, Fujita M. Building a database for brain 18 kDa translocator protein imaged using [11C]PBR28 in healthy subjects. J Cereb Blood Flow Metab. 2019 Jun;39(6):1138-1147. doi: 10.1177/0271678X18771250. Epub 2018 May 11. PMID 29749279
- [Derived] Kreisl WC, Lyoo CH, Liow JS, Snow J, Page E, Jenko KJ, Morse CL, Zoghbi SS, Pike VW, Turner RS, Innis RB. Distinct patterns of increased translocator protein in posterior cortical atrophy and amnestic Alzheimer's disease. Neurobiol Aging. 2017 Mar;51:132-140. doi: 10.1016/j.neurobiolaging.2016.12.006. Epub 2016 Dec 16. PMID 28068564
- [Derived] Kreisl WC, Lyoo CH, Liow JS, Wei M, Snow J, Page E, Jenko KJ, Morse CL, Zoghbi SS, Pike VW, Turner RS, Innis RB. (11)C-PBR28 binding to translocator protein increases with progression of Alzheimer's disease. Neurobiol Aging. 2016 Aug;44:53-61. doi: 10.1016/j.neurobiolaging.2016.04.011. Epub 2016 Apr 27. PMID 27318133
- [Derived] Lyoo CH, Ikawa M, Liow JS, Zoghbi SS, Morse CL, Pike VW, Fujita M, Innis RB, Kreisl WC. Cerebellum Can Serve As a Pseudo-Reference Region in Alzheimer Disease to Detect Neuroinflammation Measured with PET Radioligand Binding to Translocator Protein. J Nucl Med. 2015 May;56(5):701-6. doi: 10.2967/jnumed.114.146027. Epub 2015 Mar 12. PMID 25766898